CLINICAL TRIAL: NCT05208424
Title: Incidence, Characteristics and Outcome of Patients With New Diabetes Mellitus and Pre-Diabetes With First-time Diagnosed Coronary Artery Disease
Brief Title: New Diabetes Mellitus and Pre-Diabetes With First-time Diagnosed Coronary Artery Disease
Acronym: DMCAD
Status: Completed | Type: Observational
Sponsor: Saud Al Babtain Cardiac Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: IRB-2020-02
Record Dates: First submitted 2021-12-23; First posted 2022-01-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: PreDiabetes; Diabetes; Coronary Artery Disease
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus; Coronary Artery Disease | interventions — Coronary Angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal glycemia: 100 patients without evidence of dysglycemia.
  Interventions: Diagnostic Test: Coronary angiography
- Prediabetes: 100 patients with evidence of pre-diabetes defined as hemoglobin A1C (HbA1c) 5.7-6.4% with or without fasting plasma glucose (FPG) of 100 mg/dL to 125 mg/dL.
  Interventions: Diagnostic Test: Coronary angiography
- Diabetes: 100 patients without evidence diabetes defined as hemoglobin HbA1c > 6.4% with or without FPG >125 mg/dL.
  Interventions: Diagnostic Test: Coronary angiography

INTERVENTIONS:
Diagnostic Test: Coronary angiography — Invasive coronary angiography

SUMMARY:
A prospective analytic study to evaluate the incidence, clinical and laboratory characteristics, extent of coronary artery disease and short-term outcome of newly diagnosed diabetes and pre-diabetes in patients with first-time diagnosed coronary artery disease treated in Saud Al Babtain Cardiac Center.

ELIGIBILITY:
Inclusion Criteria:

* First time diagnosed coronary artery disease as confirmed by invasive coronary angiography
* Emergently or electively admitted as coronary artery disease patients.
* Informed consent form

Exclusion Criteria:

* Prior diagnosis of diabetes or pre-diabetes based on the diagnostic criteria of the American Diabetes Association (ADA, 2020)
* Known coronary artery disease

Min Age: 18 Months | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients with first time diagnosed coronary artery disease, based on invasive coronary angiography, with no prior history of dysglycemia will be enrolled from all comers to Saud AlBabtain Cardiac Center
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence | Through study completion, an average of 2 year
  The incidence, number and percent, of newly diagnosed diabetes and pre-diabetes in patients with first-time diagnosed coronary artery disease
Characteristics, clinical and laboratory | Through study completion, an average of 2 year
  Clinical and laboratory characteristics of newly diagnosed diabetes and pre-diabetes in Patients with first-time diagnosed coronary artery disease.
Coronary artery disease severity | Through study completion, an average of 2 year
  Extent of newly diagnosed coronary artery disease in newly diagnosed diabetes and pre-diabetes. The severity of coronary artery disease will be assessed using the SYNTAX score.
Short-term outcome | From admission to 1-month follow up.
  Assessment will include in-hospital and 1-month major adverse cardiac events (MACE), recurrent angina, stent thrombosis, need for emergent/urgent coronary intervention, clinical heart failure and left ventricular dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- Saud AlBabtain Cardiac Center, Dammam, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Diabetes Association. 2. Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2021. Diabetes Care. 2021 Jan;44(Suppl 1):S15-S33. doi: 10.2337/dc21-S002. PMID 33298413
- [Background] Zhang YJ, Iqbal J, Campos CM, Klaveren DV, Bourantas CV, Dawkins KD, Banning AP, Escaned J, de Vries T, Morel MA, Farooq V, Onuma Y, Garcia-Garcia HM, Stone GW, Steyerberg EW, Mohr FW, Serruys PW. Prognostic value of site SYNTAX score and rationale for combining anatomic and clinical factors in decision making: insights from the SYNTAX trial. J Am Coll Cardiol. 2014 Aug 5;64(5):423-32. doi: 10.1016/j.jacc.2014.05.022. PMID 25082573